Official Title: A Phase IIA, International, Multicenter, Open-Label, Uncontrolled

Study to Evaluate the Safety and Pharmacokinetics of  $4\times375$  mg/m2 Intravenous Rituximab in Pediatric Patients With Severe Granulomatosis With Polyangiitis (Wegener's) or Microscopic

**Polyangiitis** 

NCT Number: NCT01750697

**Document Date:** Data Analysis Plan, Module 2, Version 1.0, dated 10-Sep-2018

### DATA ANALYSIS PLAN - MODULE 2

TITLE:

A PHASE IIa, INTERNATIONAL, MULTICENTER, OPEN-LABEL, UNCONTROLLED STUDY TO EVALUATE THE SAFETY AND PHARMACOKINETICS OF 4 × 375 mg/m<sup>2</sup> INTRAVENOUS RITUXIMAB IN PEDIATRIC PATIENTS WITH

SEVERE GRANULOMATOSIS WITH POLYANGIITIS (WEGENER'S) OR MICROSCOPIC POLYANGIITIS

PROTOCOL NUMBER:

WA25615

STUDY DRUG:

Rituximab (RO0452294)

SPONSOR:

Author:

F. Hoffmann-La Roche Ltd for 1.0

**VERSION NUMBER:** 

Approver:

This is a F. Hoffmann-La Roche Ltd document that contains confidential information. Nothing herein is to be disclosed without written consent from F. Hoffmann-La Roche Ltd.

Rituximab-F. Hoffmann-La Roche Ltd.

WA25615: DAP Module 2

<sup>\*</sup> The approver has ensured that key team members have been involved, contributed and reviewed the content of the List of Planned Outputs as described in the DAP Module 2 guideline.

### **TABLE OF CONTENTS**

| 1. | BACKGRO | OUND | 4 |
|---|---|---|---|
| 2. | STUDY DESIGN | | |
| | 2.1 | Outcome Measures | 5 |
| | 2.1.1 | Primary Safety Outcome Measures | 5 |
| | 2.1.2 | Primary Pharmacokinetic Outcome Measures | 5 |
| | 2.1.3 | Secondary Pharmacokinetic Outcome Measures | 5 |
| | 2.1.4 | Primary and Secondary Efficacy Outcome Measures | 5 |
| | 2.1.5 | Secondary Safety Outcome Measures | 5 |
| | 2.1.6 | Exploratory Outcome Measures | 6 |
| | 2.1.6 | 6.1 Exploratory Efficacy Outcome Measures | 6 |
| | 2.1.6 | 5.2 Exploratory Pharmacodynamic Outcome Measures | 9 |
| | 2.2 | Determination of Sample Size | 9 |
| | 2.3 | Analysis Timing | 9 |
| | 2.3.1 | Data Included in the Remission Induction Phase | 9 |
| | 2.3.2 | Data Included in the Follow-up Phase | 10 |
| | 2.3.3 | Data Included in the Extended Follow-up Phase | 10 |
| 3. | STATISTICAL METHODS OVERVIEW1 | | |
| | 3.1 | Analysis Populations | 11 |
| | 3.1.1 | Safety Population | 11 |
| | 3.2 | Baseline Demographics and Baseline Information | 11 |
| | 3.2.1 | Definition of Remission Induction Phase Baseline | 11 |
| | 3.2.2 | Follow-up Phase Baseline | 11 |
| | 3.2.3 | Extended Follow-up Phase Baseline | 11 |
| | 3.3 | Visit Windows | 12 |
| | 3.4 | Analysis Overview | 13 |
| 4. | BASELINE | DEMOGRAPHICS AND BASELINE INFORMATION | 14 |
| | 4.1 | Analysis of Study Conduct | 14 |
| | 4.2 | Analysis Populations and Disposition | 15 |
| | 4.3 | Baseline Output Specifications | 15 |
| 5. | EXPOSUR | RE TO STUDY MEDICATION | 29 |
| | 5.1 | Exposure Output Specifications | 29 |

| 6. | ADVERS | SE EVENTS | 41 |
|-----|----------------------------|--------------------------------------|----|
| | Adverse | Event Output Specifications | 42 |
| 7. | SAFETY LABORATORY ANALYSES | | 50 |
| | 7.1 | Safety Laboratory Analyses | 50 |
| | 7.2 | Acute-phase Reactants | 50 |
| | 7.3 | Immunologic and Antibody Assessments | 50 |
| | 7.4 | Laboratory Output Specifications | 51 |
| 8. | VITAL SI | IGNS OUTPUT SPECIFICATIONS | 58 |
| | 8.1 | Vital Signs Output Specifications | 58 |
| 9. | EFFICAC | CY ANALYSES | 62 |
| | 9.1 | Efficacy Output Specifications | 64 |
| 10. | PHARMA | ACODYNAMIC ANALYSES | 81 |
| LIS | T OF TAB | BLES | |
| Tab | le 1 | Analysis Visit Time-point Windows | 12 |
| LIS | T OF APP | PENDICES | |
| App | endix 1 | Study Design | 94 |
| App | endix 2 | Schedule of Assessments | 95 |

### 1. BACKGROUND

This document provides specifications for the primary analysis including, remission induction phase, follow-up phase and extended follow-up phase, of the study WA25615.

- Remission Induction Phase: Day 1 until end of month 6.
- Follow-Up Phase: Post month 6 until common closeout date, where common closeout date is 18 months after the enrolment of the last patient.
- Extended Follow-Up Phase: Post common closeout date until CD19 B-cell counts have returned to baseline level or within normal range, whichever is lower.

### 2. STUDY DESIGN

This is a Phase IIa, international, multicenter, open-label, single-arm study. The primary objectives are to evaluate the safety and tolerability and the PK parameters of rituximab in pediatric patients with severe GPA or MPA.

The study comprises an initial 6-month remission induction phase; rituximab is administered on Days 1, 8, 15 and 22 during this phase. The remission induction phase is followed by a minimum 12-month follow-up phase, after which patients are followed up 3-monthly until the common closeout date, which occurs when the final participant enrolled has completed his or her Month 18 study visit (see Appendix 2).

Following the remission induction phase (month 6), if required for the maintenance of remission, further courses of rituximab may be given, with the dose and the frequency of retreatment at the discretion of the investigator.

At the common closeout date, patients whose B cells remain depleted and/or have immunoglobulin levels below the LLN for the population, continue to attend study visits every 3 months until their B-cell counts have returned to baseline level or to within the normal range for the population, whichever is lower, and until their immunoglobulin levels have returned to within normal limits for the population. Patients that receive any B-cell therapy or other agent that affects the return of B-cells including but not limited to rituximab, CYC, AZA, on or after the common closeout date, he or she will not be followed any further.

The Study Schema is given in Appendix 1 and the Schedule of Assessments is given in Appendix 2.

### 2.1 Outcome Measures

This section lists all of the study outcome measures that will be included in this analysis.

### 2.1.1 Primary Safety Outcome Measures

The primary safety outcome measures are:

- Frequency, nature, and severity of AEs
- Frequency of laboratory abnormalities

### 2.1.2 Primary Pharmacokinetic Outcome Measures

The primary PK parameters are:

• Clearance (CL) and volume of distribution

### 2.1.3 <u>Secondary Pharmacokinetic Outcome Measures</u>

The secondary PK parameters of interest are:

• AUC<sub>0-inf</sub> and C<sub>max</sub>, derived from the primary PK parameters

### 2.1.4 Primary and Secondary Efficacy Outcome Measures

None

### 2.1.5 Secondary Safety Outcome Measures

The secondary safety outcome measures are:

Vital signs

Rituximab—F. Hoffmann-La Roche Ltd

WA25615: DAP Module 2

- Electrocardiograms new or worsened abnormalities are reported as adverse events
- Chest x-ray and computed tomography (CT) scan to be completed at month 1 if abnormal at baseline and as indicated otherwise at the discretion of the investigator. New or worsened abnormalities are reported as adverse events
- Physical examinations post-baseline examinations are to be symptom directed only, with new or worsened abnormalities reported as adverse events
- Laboratory parameters (clinically relevant new or worsened abnormalities are reported as adverse events):
  - Hematology: hemoglobin, hematocrit, red blood cells and indices (mean corpuscular volume, mean cell hemoglobin, mean corpuscular hemoglobin concentration), white blood cells, absolute differential, and platelet counts
  - Serum chemistry: AST/SGOT, ALT/SGPT, alkaline phosphatase, total protein, total bilirubin (direct and indirect if total bilirubin is greater than the ULN), urea, uric acid, creatinine, potassium, sodium, chloride, calcium, phosphate, and glycosylated hemoglobin (HbA1c)
  - o Acute-phase reactants: erythrocyte sedimentation rate and C-reactive protein
  - o Urinalysis: dipstick for blood, protein, and glucose, and albumin to creatinine ratio
    - microscopic examination if abnormal and applicable
- Immunologic Assessments
  - B- and T-cell populations by fluorescence-activated cell sorter (FACS) analysis, including, but not limited to, CD3, CD4, CD8, CD16/56, CD19, CD27, CD4/45RA/45RO and CD8/45RA/45RO
  - Quantitative immunoglobulin levels (including total immunoglobulin, immunoglobulin A [IgA], IgG, and IgM isotype levels)

### 2.1.6 Exploratory Outcome Measures

# 2.1.6.1 Exploratory Efficacy Outcome Measures







### 2.2 Determination of Sample Size

The planned sample size of 25 patients was determined on the basis of the epidemiology of pediatric GPA and MPA plus information from existing patient cohorts. This sample size takes into the account the number of pediatric patients that would be eligible for treatment with rituximab and that could be expected to be enrolled within a reasonable timeframe. The primary objective of this study is to evaluate the safety and pharmacokinetics of rituximab in these patients. The planned sample size would be sufficient to provide a reasonable estimate of variability for the mean PK parameters based on the observed intra-patient variability from the RAVE study (a rituximab in ANCA-associated vasculitis trial), protocol number ITN021AI. It would also ensure 95% probability of observing at least one AE when the underlying incidence of that event is ≥11%.

Given the exploratory nature of this study, there will be no formal statistical hypothesis testing. The study will focus on exploratory estimation of the efficacy and PD endpoints.

### 2.3 Analysis Timing

There is an interim analysis for this study where the study data for the remission induction phase (6-month time-point) is analyzed when the last patient has reached the 6 month visit and the data have been cleaned with the relevant parts of the database locked for editing.

Primary analysis will be done once all of the data, up until the follow-up visit subsequent to the common closeout date (the Withdrawal visit), has been entered into the study database, cleaned and the database locked for editing.

A final analysis will be reported once the extended follow-up for all appropriate patients has been completed, with all data entered into the database, cleaned and the database fully locked.

### 2.3.1 <u>Data Included in the Remission Induction Phase</u>

The following data will be included in the analysis of the 6-month time-point:

### • Patients entering the follow-up phase:

 All screening and post-baseline data with a clinical date (i.e., administration/ assessment/onset/start date) on or before the date of entry into the follow-up phase at Month 6 will be included.

The only exceptions to this is:

 Concomitant medications that begin on the date of entry to the follow-up phase will not be included.

### • Patients not entering the follow-up phase:

All screening and post-baseline data with a clinical date on or before the date of the patient's last study visit within Study Day 210 will be included; (Day 210 equals 180 days plus a 30-day window).

The data cut will include all data regardless of the type of study visit at which it was collected. This may include data collected at unscheduled visits, dosing termination visits, early termination visits, or safety follow-up visits, if the visit date was on or before the data cutoff date.

### 2.3.2 <u>Data Included in the Follow-up Phase</u>

For patients who enter the Follow-up phase all of their screening data plus post Month-6 data with a clinical date on or before the date of entry into the Extended Follow-up Phase will be included in this analysis of the Follow-up phase.

### • Patients entering the extended follow-up phase:

All screening and post-Month-6 data with a clinical date on or before the date of entry into the extended follow-up phase will be included.

### Patients not entering the extended follow-up phase:

All screening and post-Month-6 data with a clinical date on or before the date of the patient's last study visit within common closeout date will be included.

### 2.3.3 Data Included in the Extended Follow-up Phase

Patients whose peripheral B cells remain depleted at the common closeout date will enter the Extended Follow-up phase. For patients who enter this phase all of their screening data plus post Follow-up phase data will be included in this analysis.



### 3. STATISTICAL METHODS OVERVIEW

As this is an open-label, single-arm study, with primary objectives regarding safety and PK there will be no formal statistical hypothesis testing.

The day of enrollment (Day 1) will be considered the day the patient receives their first infusion, or part thereof, of rituximab.

For binary endpoints the number and percentage of patients will be presented by visit. At key time points (Month 6, 12 and 18) two-sided 95% Confidence intervals (CIs) for the percentage of patients will be calculated.

For continuous endpoints, the n, mean, median, standard deviation (SD), minimum and maximum values will be presented by visit with two-sided 95% Cls for the mean presented for the data at key time-points (Months 6, 12 and 18), unless stated otherwise.

When we have 0 counts, please don't display 0.0%

### 3.1 Analysis Populations

### 3.1.1 Safety Population

All patients who received at least part of one infusion of rituximab will be included in the safety population.

Safety and efficacy analyses will be based on the safety population.

### 3.2 Baseline Demographics and Baseline Information

Details of the analyses and outputs are given in Section 4.

### 3.2.1 Definition of Remission Induction Phase Baseline

Baseline will be defined as the last available pre-treatment value taken on or before the initiation of rituximab (RTX) treatment on study treatment Day 1, and will be used for summary of demographic characteristics, as well as for all change-from-baseline analyses of efficacy, safety, and PD endpoints.

Special rules apply for the determination of the PVDI baseline score to account for missing individual scores: see Section 10.

For endpoints that are defined in terms of change from baseline, patients who do not have a pretreatment value reported for a particular assessment (if any) will be excluded from the change-frombaseline analyses for that assessment.

### 3.2.2 Follow-up Phase Baseline

The Follow-up phase will use the same baseline values as the Remission Induction phase for all analyses.

### 3.2.3 Extended Follow-up Phase Baseline

Baseline will be defined as the last available value taken on or before the start of the Extended Follow-up phase, and will be used for all change-from-baseline analyses of safety and PD

endpoints. For B cell deplection (absolute CD19 count) we should use the baseline value prior to receiving study medication.

For endpoints that are defined in terms of change from baseline, patients who do not have a pretreatment value reported for a particular assessment (if any) will be excluded from the change-frombaseline analyses for that assessment.

### 3.3 Visit Windows

For summarization by time-point data will be assigned to an analysis visit based on the date of the assessment relative to the date of study treatment Day 1 (treatment start). The visit assessment windows given in Table 1 will be used to assign data to planned study assessments:

| Table 1 | Analysis | Visit Time- | point Windows |
|---------|----------|-------------|---------------|
|---------|----------|-------------|---------------|

| Assessment<br>Month | Planned<br>Treatment Day (1) | Day Number (1)<br>Range |
|---|---|---|
| Baseline | 1 | Day 1 |
| Week 1 | 8 | Days 5 – 11 |
| Week 2 | 15 | Days 12 – 18 |
| Week 3 | 22 | Days 19 – 25 |
| Month 1 | 29 | Days 26 – 44 |
| Month 2 | 60 | Days 45 – 75 |
| Month 4 | 120 | Days 105 – 135 |
| Month 6 | 180 | Days 165 – 210 |
| Month 9 | 270 | Days 240 – 300 |
| Month 12 | 365 | Days 335 – 395 |
| Month 15 | 455 | Days 425 – 485 |
| Month 18 | 545 | Days 500 – 590 |
| Month 21<br>or<br>Follow-up<br>month 3 | ** | Planned<br>Treatment Day ±<br>45 days |
| Month 24<br>or<br>Follow-up<br>month 6 | ** | Planned<br>Treatment Day ±<br>45 days |

<sup>\*\*</sup> Planned Treatment Day = Month 18 Planned Treatment Day + 92 × (number of follow-up month /3)

Assessments made outside of these assessment windows will be listed but not used in *by time-point* summaries.

<sup>(1)</sup> For each patient, the day of the baseline visit will be defined as treatment day 1 and subsequent time-points will be assigned a treatment day calculated as:

(date of assessment – date of baseline) + 1

For a given measurement and analysis visit the following rules will be used to decide which value to use in the analysis:

- Protocol defined visit assessments will take priority over unscheduled visit data; that is, unscheduled visit data will only be used if there is no scheduled visit results within the same time window.
- If more than one assessment falls within the same window, then use the measurement taken nearest to the planned day. In the case of a tie, use the earlier measurement.
- Assessments made outside of these analysis visit windows will be listed but not used in by timepoint summaries.

### 3.4 Analysis Overview

### Safety Analyses

All safety analyses will be done on safety population and by study phase.

Abnormal electrocardiogram (ECG), chest X-ray and chest CT scan findings are to be reported.

Details of the analyses and outputs are given in Section  $\underline{5}$  to  $\underline{9}$ .

### Efficacy Analysis

### Pharmacodynamic Analyses

### **Subgroup Analyses**

The sample size for this study is too small to permit subgroup analyses.

### 4. BASELINE DEMOGRAPHICS AND BASELINE INFORMATION

Descriptive summaries of the following information will be produced to characterize baseline characteristics for the safety population:

- Demographic characteristics, including:
  - age, both as descriptive summary and as counts and percentages falling into the following categories:
    - 2 11 years
    - 12 17 years
  - o sex
  - o race
  - ethnicity
  - o height
  - o weight
  - o body surface area
- Baseline disease characteristics:
  - GPA or MPA disease
    - ANCA result (C-ANCA, P-ANCA, Negative)
  - o Duration of disease
  - Pediatric Vasculitis Damage Index (PVDI)
- · Previous and current treatment for GPA or MPA
  - A glossary showing the mapping of investigator verbatim terms to coded medications will be produced also
- Immunization history
- · Patients' medical history, grouped by preferred term within SOC
  - A glossary showing the mapping of investigator verbatim terms to coded diseases will be produced also
- Alcohol, tobacco and substance use
- · Female reproductive status

### 4.1 Analysis of Study Conduct

The following data will be summarized for the safety population, giving the number and percentage of patients who:

- Had major protocol deviations occurring during the remission induction phase
- Were withdrawn prematurely from the study
- Entered extended follow-up (To be added later as CSR addendum)
- Entered extended follow-up
- Switched to local standard care during the study by study phase

In addition, summaries will be provided of:

- Non-study treatments given for GPA and MPA by study phase
- · Concomitant medications received by study phase

### 4.2 Analysis Populations and Disposition

The following summaries will be produced:

- · Analysis populations
- Patient disposition by study phase (remission induction phase, follow-up phase, extended follow-up phase)

### 4.3 Baseline Output Specifications

| ID: DS101SP | STREAM Template: APT01 |
|---|---|
| Analysis Populations | |
| | <b>Analysis Variables:</b> Number of patients for the only analysis population, as shown in the mockup. |
| | Numeric Precision and Formatting of Statistics: Use mockup. |

| Analysis Population | Rituximab |
|---|---|
| Treated Patients AASL.RP (Assigned Treatment AASL.ARM) | nn |
| Safety Evaluable Population ASL.SE (Treatment Received AASL.ACTARM) | nn (xx.x%) |
| Population (Safety population with at least one evaluable PK sample) | nn (xx.x%) |

## ID: DS001SP Enrolment by Region, Country, and Investigator Number and Name STREAM Template: ENT02 Analysis Population: Samedical history fety Evaluable Population Analysis Variables: Group centers by region and country. Sort order: Alphabetical by region, and then by decreasing total number of patients treated. Percentages are based on N. Numeric Precision and Formatting of Statistics: Use standard display in the mockup.

| Region ASL.GEOREGC1 Country ASL.COUNTRY, Investigator Number ASL.INVID / Name ASL.INVNAM | Rituximab<br>(N=nnn) |
|---|---|
| Region 1 | nn (xx.x%) |
| Country 1 | nn (xx.x%) |
| 9318 / Name 1 | nn (xx.x%) |
| 11518 / Name 2 | nn (xx.x%) |
| | nn (xx.x%) |
| Country 2 | nn (xx.x%) |
| 88431 / Name 1 | nn (xx.x%) |
| 8876 / Name 2 | nn (xx.x%) |
| | nn (xx.x%) |
| Region 2 | nn (xx.x%) |
| Country 1 | nn (xx.x%) |
| 77649 / Name 1 | nn (xx.x%) |
| | nn (xx.x%) |

| ID: DM001SP | STREAM Template: DMT01 |
|---|---|
| Demographic and<br>Baseline Characteristics | Analysis Population: Safety Evaluable Population |
| | Analysis Variables: See mockup. |
| | Statistics and Calculation Methods: For each variable, summary statistics are based on the number of patients in the corresponding "n" row. |
| | Number of concomitant diseases started before or at baseline and continued after. |
| | Numeric Precision and Formatting of Statistics: Use standard display in the mockup. |

| | Rituximab<br>(N=nnn) |
|----------------------------------|--------------------------|
| Age (yr) ASL.AGE | (** *****) |
| n | nnn |
| Mean (SD) | xx.x (xx.x) |
| Median | XX.X |
| Q1 – Q3 (IQR) | xx.x - xx.x (xx.x) |
| Min-Max | XX-XX |
| Age group (yr) ASL.AGEG | |
| n | nnn |
| 2 to 11 | nn (xx.x%) |
| 12 to 17 | nn (xx.x%) |
| 0 401 0TV | |
| Sex ASL.SEX | nnn |
| n<br>Male | nnn |
| Female | nn (xx.x%)<br>nn (xx.x%) |
| remale | IIII (XX.X70) |
| Ethnicity ASL.ETHNIC | |
| n ´ | nnn |
| Hispanic or Latino | nn (xx.x%) |
| Not Hispanic or Latino | nn (xx.x%) |
| Not Reported | nn (xx.x%) |
| Unknown | nn (xx.x%) |
| Race ASL.RACE | |
| n | nnn |
| American Indian or Alaska Native | nn (xx.x%) |
| Asian | nn (xx.x%) |
| Black or African American | nn (xx.x%) |
| Native Hawaiian or | nn (xx.x%) |
| other Pacific Islander | ···· (/du///d |
| White | nn (xx.x%) |
| Multiple | nn (xx.x%) |
| Other | nn (xx.x%) |
| Unknown | nn (xx.x%) |
| Height (cm) ASL.BWT | |
| n<br>Maan (CD) | nnn |
| Mean (SD) | xx.x (xx.x) |
| Median | XX.X |
| Q1 – Q3 (IQR)<br>Min–Max | xx.x - xx.x (xx.x) |
| IVIII I—IVI <b>a</b> X | XX–XX |

| | Rituximab<br>(N=nnn) |
|---|---|
| Weight (kg) ASL.BWT | , , |
| n S | nn |
| Mean (SD) | XX.X (XX.X) |
| Median | XX.X |
| Q1 – Q3 (IQR) | xx.x - xx.x (xx.x) |
| Min-Max | XX-XX |
| THIS THEAT | AA AA |
| Body-mass index (kg/m2) ASL.BBMI | |
| n<br>M (OD) | nn |
| Mean (SD) | xx.x (xx.x) |
| Median | XX.X |
| Q1 – Q3 (IQR) | xx.x - xx.x (xx.x) |
| Min-Max | XX-XX |
| Concomitant Diseases (continuing at Baseline) | |
| n | nn |
| No concomitant diseases | nn (xx.x%) |
| 1 concomitant disease | nn (xx.x%) |
| 2 concomitant diseases | nn (xx.x%) |
| >=3 concomitant diseases | nn (xx.x%) |
| 7-0 concomitant diseases | 1111 (22.270) |
| Smoking history | |
| n | nn |
| Current | nn (xx.x%) |
| Previous | nn (xx.x%) |
| Never | nn (xx.x%) |
| Alcohol history n Current Previous Never | nn<br>nn (xx.x%)<br>nn (xx.x%)<br>nn (xx.x%) |
| Estimated GFR (Schwartz formula) (mL/min/1.73 m2) n Mean (SD) Median | nn<br>xx.x (xx.x)<br>xx.x |
| Q1 – Q3 (IQR) | xx.x - xx.x (xx.x) |
| Min-Max | XX.X-XX.X |
| immunofluorescence (IF) ANCA | |
| status | |
| Negative | nn (xx.x%) |
| cANCA | nn (xx.x%) |
| pANCA | nn (xx.x%) |
| MPO | nn (xx.x%) |
| PR3 | nn (xx.x%) |
| | IIII (AA.A70) |
| BVAS/WG Score<br>n | nn |
| Mean (SD) | xx.x (xx.x) |
| Median | XX.X |
| Q1 – Q3 (IQR) | xx.x - xx.x (xx.x) |
| Min-Max | XX.X-XX.X |

```
Current Disease Status
   Severe Flare/New Disease
                                               nn (xx.x%)
   Limited Flare/New Disease
                                               nn (xx.x%)
   Persistent Severe Disease
                                               nn (xx.x%)
   Persistent Limited Disease
                                               nn (xx.x%)
   Remission
                                               nn (xx.x%)
BVAS/WG PGA
                                                   nn
   Mean (SD)
                                               xx.x (xx.x)
   Median
                                                  XX.X
   Q1 - Q3 (IQR)
                                            XX.X - XX.X (XX.X)
   Min-Max
                                               XX.X-XX.X
PVAS Score
                                                  nn
   Mean (SD)
                                               XX.X (XX.X)
   Median
                                                  XX.X
   Q1 - Q3 (IQR)
                                            XX.X - XX.X(XX.X)
   Min-Max
                                               XX.X-XX.X
PVDI Score
                                                   nn
   Mean (SD)
                                               xx.x (xx.x)
   Median
                                                  XX.X
   Q1 - Q3 (IQR)
                                            XX.X - XX.X (XX.X)
   Min-Max
                                               XX.X-XX.X
PVDI Average School Absence (days)
                                                   nn
   =<1
                                               nn (xx.x%)
   >1 - 4
                                               nn (xx.x%)
   >4 - 10
                                               nn (xx.x%)
   >10
                                               nn (xx.x%)
```

| ID: DM002SP | STREAM Template: DMT01 |
|---|---|
| GPA / MPA History | Analysis Population: Safety Evaluable Population |
| | Analysis Variables: See mockup. |
| | Statistics and Calculation Methods: For each variable, summary statistics are based on the number of patients in the corresponding "n" row. |
| | Major Renal Disease is taken from eCRF page, BVAS/ WG and PGA. If both hematuria and RBC casts are present, score only the RBC casts. |
| | Summaries are based on Medical history and Concomitant medication domains, and Screening records for other assessments. |
| | Most severe "Current Disease Status" is used for summary if patient has multiple disease status from Screening. |
| | Disease duration is from the start date of disease to start of study drug at baseline. |
| | Numeric Precision and Formatting of Statistics: See mockup. |

| | Rituximab<br>(N=nnn) |
|---|---|
| Diagnosis | |
| n<br>GPA Newly diagnosed<br>MPA Newly diagnosed<br>GPA relapsed<br>MPA relapsed | nn<br>nn (xx.x%)<br>nn (xx.x%)<br>nn (xx.x%)<br>nn (xx.x%) |
| Disease duration (months) n Mean (SD) Median Q1 – Q3 (IQR) Min–Max | nn<br>xx.x (xx.x)<br>xx.x<br>xx.x – xx.x (xx.x)<br>xx–xx |
| Prior CYC therapy | |
| n<br>Yes<br>No | nn<br>nn (xx.x%)<br>nn (xx.x%) |
| Major Renal Disease* n Yes No | nn<br>nn (xx.x%)<br>nn (xx.x%) |

<sup>\*</sup> Major Renal Disease is taken from eCRF page, BVAS/ WG and PGA. If both hematuria and RBC casts are present, score only the RBC casts (the major item)









| ID: DM003SP | STREAM Template: DSL02 |
|---|---|
| Listing of Patients who | Analysis Population: Safety Evaluable Population |
| Discontinued from<br>Study | Variables Displayed: Add a columns for "date of study discontinuation" and "study phase" to DSL02 |

| ID: DS201SP | STREAM Template: DST01 |
|---------------------|--------------------------------------------------|
| Patient Disposition | Analysis Population: Safety Evaluable Population |
| - | Analysis Variables: See mockup. |

| Study | Rituximab |
|---------------------------------------------------|-------------|
| | (N = 25) |
| Completed 6 Month Remission Induction Phase | nn (xx.xx%) |
| Completed 18 Months on study | nn (xx.xx%) |
| Completed study from baseline to common-closeout* | nn (xx.xx%) |
| Entered extended safety follow-up+ | nn (xx.xx%) |
| Discontinued Study | nn (xx.xx%) |
| Reason 1 | nn (xx.xx%) |
| Reason 2 | nn (xx.xx%) |
| Reason 3 | nn (xx.xx%) |

<sup>\*</sup>The common closeout date (10May2018) occurred 18 months after the enrollment of the last patient.
+patients whose B cells remain depleted below LLN for the population entered extended safety follow up.

| ID: DS002SP | STREAM Template: DST01 |
|---|---|
| Patients Discontinued | Analysis Population: Safety Evaluable Population |
| from Study Treatment | Analysis Variables: See mockup |

| Status | | uximab<br>=25) |
|---|---|---|
| Completed Planned RTX Treatment Discontinued Treatment During Study Lost To Follow-Up Patient Is Transitioning To Adult Care. Transfer To Adult Services Transfered To Adult Services And Upable To Stay In Follow Up Of P Transferred To Adult Site Transferring To Adult Services Withdrawal By Subject | nn<br>nn<br>nn<br>nn<br>i nn<br>nn<br>nn | (xx.x%) |

| ID: CM001SP | STREAM Template: None |
|---|---|
| Listing of Concomitant | Analysis Population: Safety Evaluable Population |
| Diseases other than<br>MPA/GPA | Variables Displayed: See mockup. |
| WINGIA | Concomitant Disease is defined as a disease started on or before baseline and continued after. |
| | Exclude MPA/GPA diseases from the listing. |

| Center/Patient ID - Age/Sex/Race<br>Concurrent Disease<br>MedDRA Preferred Term | Date of First<br>Study Drug<br>Administration | Start Date of Disease<br>/ Study Day of onset | Duration<br>in Days | Outcome |
|---|---|---|---|---|
| ANEAMIA NOS APPETITE DECREASED | | / -60<br>/ -91 | 1 2 | Resolved<br>Resolved |
| DIARRHEA NOS | | / -425 | 2 | Resolved |

| ID: CM002SP | STREAM Template: None |
|---|---|
| Listing of Previous | Analysis Population: Safety Evaluable Population |
| Medications for<br>GPA/MPA | Variables Displayed: Include medications started and ended on or before baseline. |
| | See mockup. |



| ID: CM003SP | STREAM Template: None |
|---|---|
| Listing of Concomitant | Analysis Population: Safety Evaluable Population |
| Medications for<br>GPA/MPA | Variables Displayed: Include medications started anytime (after, on or before baseline) and is ongoing during study. |
| | See mockup. |

| Center/Patient ID - Age/Sex/Race<br>Standardized Medication Name<br>Reported Name of Drug,<br>Medication or Therapy | Dose<br>(unit) | Date of First<br>Study Drug<br>Administration | Start Date of<br>Concomitant<br>Medication / Study<br>Day | Stop Date of<br>Concomitant<br>Medication / Study<br>Day |
|---|---|---|---|---|
| ANEAMIA NOS | XX | | / -34 | -34 |
| APPETITE<br>DECREASED | XX | | / -122 | / -122 |
| | XX | | | |
| DIARRHEA NOS | | | / -78 | / -78 |

1446

### ID: CM003.1SP Listing of Concomitant Medications for GPA/MPA Ongoing at Baseline STREAM Template: None Analysis Population: Safety Evaluable Population Variables Displayed: Include medications started on or before baseline and is ongoing at baseline. See mockup CM003SP.

| ID: CM003.2SP | STREAM Template: None |
|---|---|
| Listing of Concomitant | Analysis Population: Safety Evaluable Population |
| Medications for non<br>GPA/MPA Indications | Variables Displayed: Include medications started anytime (after, on or before baseline) and is ongoing during study for non MPA/GPA indications. |
| | Exclude vaccines from the con meds if the start date is before day 1. |
| | See mockup for CM003SP. |

| ID: MH001SP | STREAM Template: DMT01 |
|---|---|
| Immunization History | Analysis Population: Safety Evaluable Population |
| , | Analysis Variables: See mockup. |
| | Statistics and Calculation Methods: For each variable, summary statistics are based on the number of patients in the corresponding "n" row. |
| | Numeric Precision and Formatting of Statistics: See mockup |

1447

| | Rituximab<br>(N=nnn) |
|---------------------------------|----------------------|
| Tetanus Immunoglobulin | |
| n | nn |
| Yes | nn (xx.x%) |
| No | nn (xx.x%) |
| Hepatitis B Immunoglobulin | |
| n | nn |
| Yes | nn (xx.x%) |
| No | nn (xx.x%) |
| Hepatitis A Immunoglobulin | |
| n | nn |
| Yes | nn (xx.x%) |
| No | nn (xx.x%) |
| Rabies Antiserum | |
| n | nn |
| Yes | nn (xx.x%) |
| No | nn (xx.x%) |
| Varicella Zoster Immunoglobulin | |
| n | nn |
| Yes | nn (xx.x%) |
| No | nn (xx.x%) |
| Other Immunoglobulin | |
| n | nn |
| Yes | nn (xx.x%) |
| No | nn (xx.x%) |

| ID: MH001_1SP | STREAM Template: DMT01 |
|---|---|
| Vaccination History | Analysis Population: Safety Evaluable Population |
| | Analysis Variables: See mockup. |
| | Statistics and Calculation Methods: For each variable, summary statistics are based on the number of patients in the corresponding "n" row. |
| | Use CMCAT = "VACCITINATOIN" and CMOCCUR='Y'. |
| | Numeric Precision and Formatting of Statistics: See mockup |

| | Rituximab<br>(N=nnn) |
|----------------------------|----------------------|
| Tetanus Immunoglobulin | nn (xx.x%) |
| Hepatitis B Immunoglobulin | nn (xx.x%) |
| Hepatitis A Immunoglobulin | nn (xx.x%) |
| Rabies Antiserum | nn (xx.x%) |

### 5. EXPOSURE TO STUDY MEDICATION

### 5.1 Exposure Output Specifications

The following data will be presented:

- Number (%) of patients receiving 1, 2, etc. infusions of RTX
- Cumulative dose of RTX by infusion number.
- Total dose, and the number of doses of methylprednisolone prior to first dose of RTX
- Oral corticosteroid treatment duration (months), summarized both descriptively and as number (%) of patients using the following duration categories:
  - Remission induction phase<sup>(1)</sup>
    - <1 month (<26 days)</p>
    - 1 month <2 months (<45 days)
    - 2 months <4 months (<105 days)</li>
    - 4 months <6 months (<165 days)</li>
    - 6 months (≥165 days)
  - o Follow-up phase
    - 6 months <12 months (<335 days)</li>
    - 12 months <18 months (<515 days)</li>
    - 18 months <2 years (<699 days)
    - 2 years <3 years (<1067 days)</li>
    - 3+ years (≥1067 days)
- Total dose of corticosteroid following first dose of RTX.
- duration (months) in the study phases over all patients, summarized as for Methylprednisolone, above
- (1) Total duration will be calculated as:
  - 1 + Study end date Date rituximab first administered

where "study end date" is defined as:

- 1. For ealy discontinuation or completion patients: early withdrawal/discontinuation date or date patient completed study
- 2. For the rest of patients: minimum of common closeout date and last known alive date

### ID: FX001SP

Rituximab Treatment Exposure by visit during Remission Induction Phase STREAM Template: None

Analysis Population: Safety Evaluable Population

Analysis Variables: Number of infusions started, Number infusions completed without them being interrupted/modified, Number of patients with interrupted/modified infusions by infusion number, total dose of RTX. The number of infusions categories need to run from 1 (0 for number completed if necessary) to the maximum number of infusions started.

Analysis visits to include are: Baseline, Weeks 1 to 3, Months 1, 2, 4, 6 **Statistics and Calculation Methods:** The Infusion Interrupted/Modified rows count the number of Yes's from the "Was the infusion interrupted/modified" question and the denominator for the %s will be the number of patients who started that infusion number and so will correspond to the appropriate row from "Number of infusions started".

Percentages are based on:

- 1. for "Infusion started" section: based on n
- 2. for "Infusion Interrupted/Modified" section: based on nn\*, where nn\* is the number of infusions in corresponding visit.

```
Rituximab
(N=nn)
Infusions started
                                   nn
                             nn* (xx.x%)
Baseline
                              nn* (xx.x%)
Week 1
Week 2
                              nn* (xx.x%)
Week 3
                              nn* (xx.x%)
                              nn* (xx.x%)
Month 1
Infusion Interrupted/Modified
                                   nn
Baseline
                              nn/nn* (xx.x%)
                              nn/nn* (xx x%)
Week 1
                              nn/nn* (xx.x%)
nn/nn* (xx.x%)
Week 2
Week 3
                              nn/nn* (xx.x%)
Month 1
Total number of infusions completed
0
                               nn (xx.x%)
1
                               nn (xx.x%)
                               nn (xx.x%)
Total cumulative dose(mg)
                                   nn
Mean (SD)
                              xxx.x (xx.x)
Median
                                   XX.X
Q1 - Q3 (IQR)
                              xx.x- xx.x (xx.x)
Min - Max
                               XX - XXX
```

### ID: EX001.1SP

Summary of Rituximab Exposure STREAM Template: None

Analysis Population: Safety Evaluable Population

**Analysis Variables:** See mock. Percentages are based on n. Include data from Day 1 to common closeout date.

- study end date =
- 1. For ealy discontinuation or completion patients: minimum of or early withdrawal/discontinuation or patient completed study
- 2. For the rest of patients: minimum of common closout date and last known alive date

Duration of observation = study end date - study start date + 1.

Date of last contact is the last available date of efficacy, complete medication start date, laboratory, adverse event assessments, early withdrawal visit, date of last contact or date of death.

```
Total number of Infusions administered
   Mean (SD)
                               xxx.x (xx.x)
   Median
                             XX.X
                             xx.x-xx.x(xx.x)
   Q1-Q3 (IQR)
   Min - Max
                                 XX - XXX
Total cumulative dose(mg)
                                    nn
   Mean (SD)
                               xxx.x (xx.x)
   Median
                       XX.X
   Q1-Q3 (IQR)
                                 xx.x-xx.x(xx.x)
   Min - Max
                                XX - XXX
Duration of Observation (Months)
   Mean (SD)
                                  xx.x (xx.x)
   Median
                                  XX.X
   Q1-Q3 (IQR)
                                xx.x-xx.x(xx.x)
   Min - Max
                                 xx.x - xx.x
Duration of Observation (Months)
                                    nn
                                   nn (xx.x%)
nn (xx.x%)
   Duration ≤ 6
   6 < Duration ≤ 12
                                   nn (xx.x%)
   12 < Duration ≤ 18
   18 < Duration ≤ 24
                                   nn (xx.x%)
   24 < Duration ≤ 36
                                   nn (xx.x%)
   36 < Duration ≤ 48
                                   nn (xx.x%)
   48 < Duration ≤ 60
                                   nn (xx.x%)
       Duration > 60
                                   nn (xx.x%)
   Total patient years of observation xxx.xx
```

Rituximab
Administration over
Course of study

STREAM Template: None

Analysis Population: Safety Evaluable Population

Plot of:
Y-Axis: Patient ID

X-Axis: Study Visit
See mockup.



### ID: EX002SP

Listing of Rituximab Administrations, Interruptions and Modifications STREAM Template: None

Analysis Population: Safety Evaluable Population

**Column Variables:** Include data from Day 1 to common closout date.

Add "Dose Administered" column in "mg/m²" calculating as follows:

administered dose (mg/m²) = dose administered (mg) / BSA (m²),

where

BSA = body surface area = sqrt [BW x Ht / 3600]

BW = weight (kg)

Ht = height (cm)

See mockup

Sorting: Sort by center / patient ID and treatment administration day.

| Center / Patient ID ASL.SITEI D/AAE.PAT NUM | Age/Sex/R<br>ace<br>ASL.AGE/<br>ASL.SEX/<br>ASL.RACE | Height<br>(cm) /<br>Weigh<br>t (kg) | Targ<br>et<br>Day | Study<br>Day | Study<br>Visit | Planned<br>Dose<br>(mg) | Dose<br>Administere<br>d<br>(mg) | Dose<br>Administe<br>red<br>(mg/m²) | Volume<br>Administe<br>red<br>(mL) | Infusion<br>Interrupted<br>/ Modified | Reason<br>for<br>Modificatio<br>n |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 1 | 1 | baseline | xxx | 478.8 | xxx | xxx | No | |
| | | | 8 | 8 | week 2 | XXX | 479.2 | XXX | XXX | No | |
| | | | 15 | 15 | week 2 | xxx | 479.2 | xxx | xxx | Yes | Medication<br>Error |
| | | | 22 | 22 | month 1 | XXX | 482.5 | xxx | xxx | No | |

### ID: EX003SP

Corticosteroid Treatment Exposure during Remission Induction Phase and Overall **STREAM Template:** EXT01

Analysis Population: Safety Evaluable Population

Analysis Variables: Oral steroids: duration of use and total dose.

All steroids (all route) total use. This needs discussing with as she has indicated that she will not be able to supply conversion factors for non-oral steroids.

Percentages are based on n.

```
Phase: ...
                                         Rituximab
                                          (N=25)
ORAL CORTICOSTEROID DRUGS
  Treatment duration (D)
                                           25
    Mean (SD)
                                      xxx.x (xx.x)
    Median
                                        XX.X
    Q1 - Q3 (IQR)
                                     xx.x - xx.x (xx.x)
    Min - Max
                                       xx - xxx
  Treatment duration
    n
                                          nn
                                       nn (xx.x%)
    <1 month (1-25 days)
    1 - <2 months (26-44 days)
                                     nn (xx.x%)
nn (xx.x%)
    2 - <4 months (45-104 days)
                                      nn (xx.x%)
    4 - <6 months (105-164 days)
    6 months (>=165 days)
                                        nn (xx.x%)
  Total cumulative oral dose(mg)
                                           nn
    Mean (SD)
                                      xxx.x (xx.x)
    Median
                                      XX.X
    <mark>Q1 - Q3 (IQR)</mark>
Min - Max
                                      xx.x - xx.x (xx.x)
xx - xxx
ALL CORTICOSTEROID DRUGS
  Total cumulative dose (mg)
    Mean (SD)
                                      xxx.x (xx.x)
    Median
                                        XX.X
                                      xx.x - xx.x (xx.x)
xx - xxx
   Q1 - Q3 (IQR)
Min - Max
```

| ID: EX004SP | STREAM Template: None |
|---|---|
| Listing of Steroid<br>Use | Analysis Population: Safety Evaluable Population |
| | Variables Displayed: See mockup. |
| | Sorting: Sort by center / patient ID and treatment administration day. |

| Center / Patient ID ASL.SITEI D/AAE.PAT NUM | Age/Sex/Race ASL.AGE/ ASL.SEX/ ASL.RACE | Height (cm) /<br>Weight (kg) | Start<br>Day | End Day | Medication | Dose<br>Administered | Unit | Route |
|---|---|---|---|---|---|---|---|---|
| | | | 1 | 1 | DEXAMETH<br>ASONE * | 8 | mg | Intrave<br>nous |
| | | | 8 | 9 | | 479.2 | | |
| | | | 15 | 15 | | 479.2 | | |
| | | | 22 | 22 | | 482.5 | | |
| | | | 1 | 1 | | 322.5 | | |
| | | | 8 | 8 | | 322.5 | | |
| | | | 15 | 15 | | 322.5 | | |

<sup>\*</sup> GPA/MPA, PRE-RITUXIMAB INFUSION AND GLUCOCORTICOID CONCOMITANT MEDICATIONS
## ID: EX006SP

Methylprednisolone Treatment Exposure During Screening Period Prior to First Rituximab Infusion STREAM Template: EXT01

Analysis Population: Safety Evaluable Population

Analusis Variables: See mockup.

Methylprednisolone (30 mg/kg, up to 1 g/day) include Methylprednisolone dose on or before Day 1

for the number of doses, include number anf percentage of patients

having 1, 2, 3 and >3 doses.

Statistics and Calculation Methods: Prcentages are based on n.

Sorting: Sort by center / patient ID and treatment administration

day.

| | Rituximab (N=nnn) |
|----------------------------|-------------------|
| Treatment duration (D) | |
| n | nn |
| Mean (SD) | xx.x (xx.x) |
| Median | xx.x |
| Q1-Q3 (IQR) | xx.x-xx.x (xx.x) |
| Min-max | xx-xx |
| Number of doses | |
| n | nn |
| 1 dose | xx.x (xx.x%) |
| 2 doses | xx.x (xx.x%) |
| 3 doses | xx.x (xx.x%) |
| > 3 doses | xx.x (xx.x%) |
| Total cumulative dose (mg) | |
| n | nn |
| Mean (SD) | xx.x (xx.x) |
| Median | XX.X |
| Q1-Q3 (IQR) | xx.x-xx.x (xx.x) |
| Min-max | XX-XX |

| ID: EX007SP | STREAM Template: None |
|---|---|
| Patient Profile of | Analysis Population: Safety Evaluable Population |
| Oral Steroid Use | Plot of: |
| | Y-Axis: Daily prednisolone equivalent dose (mg) |
| | X-Axis: Study Visit |
| | One plot for each patient. |
| | <b>Reference lines:</b> Draw reference lines through the x-axis on the days of RTX administration. |

# Patient Profile of Oral Steroid Use, Safety-Evaluable Patients Protocol: WA25615



# ID: EX007.1SP

Patient Profiles of Cumulative Glucocorticoid Use STREAM Template: None

Analysis Population: Safety Evaluable Population

Analysis Variables: Cumulative steroid (Oral and other types in one plot with different shapes/colors) use to Months Weeks 1 to 3 and Months 1, 2, 4, 6, 12 and 18.

#### Plot of:

**Y-Axis**: Cumulative prednisone equivalent dose (mg) to time-points given above.

X-Axis: Study Visit

One plot for each patient.

Reference lines: Draw reference lines through the x-axis on the days

of RTX administration.

Numeric Precision and Formatting of Statistics: see mockup.

# Patient Profiles of Cumulative Oral Glucocorticoid Use, Safety-Evaluable Patients Protocol: WA25615



## ID: EX007.2SP

Median Glucocorticoid Use Over Time STREAM Template: None

Analysis Population: Safety Evaluable Population

Analysis Variables: Median overall steroid use (Oral and other types in two separate plots in one output file) to Weeks 1 to 3 and Months 1, 2, 4, 6, 12 and 18.

For IV, include screening period (day -28 to day 1) in the graph.

#### Plot of:

**Y-Axis**: Median overall prednisone equivalent dose (mg) to time-points given above.

X-Axis: Study Visit Error Bars: Q1 and Q3.

Numeric Precision and Formatting of Statistics: see mockup.





#### ID: EX007.3SP

Glucocorticoid Use by Visit

STREAM Template: None

Analysis Population: Safety Evaluable Population

Analysis Variables: Glucocorticoid use to Screening, Weeks 1 to 3

and Months 1, 2, 4, 6, 12 and 18.

Numeric Precision and Formatting of Statistics: see mockup.

Rituximab—F. Hoffmann-La Roche Ltd WA25615: DAP Module 2

39

| Visit | | Value at ∀isit |
|-----------|---------------|-----------------------|
| | n | nn |
| Screening | Median | xx.xx |
| | Q1 – Q3 (IQR) | xx.xx – xx.xx (xx.xx) |
| | Min - Max | XX.X - XX.X |
| Week 1 | n | nn |
| | Median | xx.xx |
| | Q1 – Q3 (IQR) | xx.xx – xx.xx (xx.xx) |
| | Min - Max | xx.x - xx.x |

### 6. ADVERSE EVENTS

Adverse events will be considered TE (defined in Section <u>4</u>) irrespective of the length of time since the first RTX infusion. Only TE adverse events will be included in summary tables. The current sponsor data safety standards will be used where available.

Summaries of TE adverse events will be produced by study phase. Summaries will be produced of the numbers of patients (%) experiencing the following TE adverse events:

Summaries will be produced of the following TE adverse events:

- Summary profile of TE adverse events
- · Overview of adverse events
- All events
- All events by most extreme toxicity grade<sup>(\*)</sup>
- Events other than IRR occurring during or within 24 hours of a RTX Infusion by relationship to treatment (count multiple occurrences as one event)
- Events leading to death
- SAEs
- SAEs assessed as related to the study drug
- Events leading to discontinuation of study medication
- Events leading to a study medication dose modification
  - o Infections
    - MedDRA SOC infections and infestations
  - Serious Infections
    - serious events in MedDRA SOC infections and infestations (include non-serious infections treated with IV anti-infective)
  - Opportunistic Infection
    - from Roche standard AEGT Opportunistic Infections
  - Infusion Related Reactions (IRRs)
    - events that occur during or within 24 hours of an infusion and fall within Roche standard AEGT Infusion Related Reactions + Hypersensitivity
    - Count multiple symptoms as one IRR for each infusion.
  - Cardiac events
    - MedDRA SOC "Cardiac Events" MedDRA SOC "Cardiac Events"
  - Malignancies
    - preferred terms in the Malignant or Unspecified Tumors SMQ (Wide)
- CTCAE grade 3 and grade 4 events
- Non-serious events reported by ≥ 5% patients (CTg requirement, not for CSR)
- Common Adverse Events reported by ≥ 10% patients

<sup>(\*)</sup> Most extreme toxicity grade is recorded on the eCRF. If most extreme toxicity grade is not recorded then initial toxicity grade will be used; if neither grade is given then an unknown category will be used. The grading is based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.

# **Adverse Event Output Specifications**

# ID: AE001SP

Overview of Adverse Events during Remission Induction Phase and Overall STREAM Template: AET01

Analysis Population: Safety Evaluable Population

Analysis Variables: See mockup

**Statistics and Calculation Methods**: Percentages are of the number of patients in SE population. For "Total number of events" rows, multiple occurrences of the same AE are counted separately. For the frequency counts by preferred term, multiple occurrences of the same AE in one individual are counted only once.

For the severe AEs (at greatest intensity), consider AEs with NCI-CTCAE grade >= 3.

Numeric Precision and Formatting of Statistics: see mockup.

| | Rituximab |
|---|---|
| | (N=nnn) |
| Total number of adverse events | nn |
| Total number of serious adverse events | nn |
| Total number of deaths | nn |
| Total number of patients with at least one | nn |
| Adverse event | nn (xx.x%) |
| Severe adverse event (at greatest intensity) | nn (xx.x%) |
| Adverse event assessed as related to study drug by investigator | nn (xx.x%) |
| Serious adverse event | nn (xx.x%) |
| Serious adverse event assessed as related to study drug by investigator | nn (xx.x%) |
| Adverse event leading to discontinuation from study treatment | nn (xx.x%) |
| Specific AEs | |
| Infection | nn (xx.x%) |
| Serious infection | nn (xx.x%) |
| Opportunistic infection | nn (xx.x%) |
| Infusion related reaction | nn (xx.x%) |
| Cardiac event | nn (xx.x%) |
| Malignancies | nn (xx.x%) |

# ID: AE002SP | STREAM Template: AET02

Adverse Events during Remission Induction Phase and Overall Analysis Population: Safety Evaluable Population

Analysis Variables: See mockup.

**Statistics and Calculation Methods**: For "Total number of AEs" rows, multiple occurrences of the same AE are counted separately. For the frequency counts by preferred term, multiple occurrences of the same AE in one individual are counted only once.

Percentages are based on N.

Numeric Precision and Formatting of Statistics: See mockup.

#### Phase: ...

| System Organ Class<br>Preferred Term | Rituximab<br>(N=25) |
|---|---|
| Overall total number of patients with at least one AE | 22 (88.0%) |
| Overall total number of AEs | 301 |
| INFECTIONS AND INFESTATIONS Total number of patients with at least one AE Total number of AEs | 16 (64.0%)<br>63 |
| UPPER RESPIRATORY TRACT INFECTION LOWER RESPIRATORY TRACT INFECTION | 10 (40.0%)<br>4 (16.0%) |

#### ID: AE002.2SP

Summary of Infusion Related Reactions (IRRs) by Visit STREAM Template: DMT01

Analysis Population: Safety Evaluable Population

Analysis Variables: See mockup.

Column Variables: Infusion numbers.

Statistics and Calculation Methods: Include two tables in one

output file:

1. For remission induction phase.

2. Foroveral period, Day 1 to common closeout date.

Infusion Related Reactions (IRRs) are defined as:

 events that occur during or within 24 hours of an infusion and fall within Roche standard AEGT Infusion Related Reactions + Hypersensitivity

Count multiple symptoms as one IRR for each infusion.

Percentages are based on n.

Visits to be included: Baseline, Week 1 to 3, month 6, 12 and 18.

Symptom of IRR = Reported term.

Numeric Precision and Formatting of Statistics: See mockup

| | Rituximab<br>(N=57) | | | | |
|---|---|---|---|---|---|
| Preferred Term/<br>Symptom of IRR | Infusion 1 | Infusion 4 | Infusion 5 | Infusion 8 | Infusion 10 |
| Number of patients who had an infusion (n) | 57 | 56 | 56 | 54 | 54 |
| Infusion related reaction* | | | | | |
| Total No. of patients with events | 5 (8.8%) | 1 (1.8%) | 2 (3.6%) | 1 (1.9%) | 0 |
| bronchospasm | 1 (1.8%) | 0 | 0 | 0 | 0 |
| cough | 1 (1.8%) | 0 | 0 | 0 | 0 |
| exanthema | 0 | 0 | 0 | 1 (1.9%) | 0 |
| metallic taste, tingling at the back of the throat | 0 | 1 (1.8%) | 0 | 0 | 0 |
| pruritus | 1 (1.8%) | 0 | 0 | 0 | 0 |
| skin rash | 1 (1.8%) | 0 | 0 | 0 | 0 |
| tightness in the throat | 0 | 0 | 1 (1.8%) | 0 | 0 |
| tingling at the back of the throat during the | 0 | 0 | 1 (1.8%) | 0 | 0 |

ID: AE004SP to

ID: AE020SP

Adverse Event Subsets during Remission Induction Phase and Overall STREAM Template: AET02

Analysis Population: Safety Evaluable Population

**Subset:** Same table contents and format, except use the following subsets (see also the beginning of this section):

| ID | Subset |
|---------|-----------------------------------------------------------------|
| AE005SP | Events resulting to death (Stream Template: AET07) |
| AE006SP | SAEs |
| AE007SP | SAEs assessed as related to the study drug |
| AE008SP | Events leading to discontinuation of study medication |
| AE009SP | Events leading to a study medication dose modification |
| AE010SP | Infections |
| | <ul> <li>MedDRA SOC infections and infestations</li> </ul> |
| AE011SP | Serious Infections |
| | <ul> <li>serious events in MedDRA SOC infections and</li> </ul> |
| | infestations |
| AE012SP | Opportunistic Infection |
| | from Roche standard AEGT Opportunistic |
| | Infections |
| AE014SP | Cardiac events |
| | MedDRA SOC "Cardiac Disorders" |
| AE015SP | Malignancies |
| | preferred terms in the Malignant or Unspecified |
| 4504000 | Tumors SMQ (Wide) |
| AE016SP | NCI CTCAE grade 3 and 4 events, using separate |
| 4504000 | sections for each grade |
| AE018SP | Events other than IRR occurring during or within 24 |
| | hours of a rituximab Infusion by relationship to |
| | treatment |

**Statistics and Calculation Methods**: Percentages are of the number of patients in SE population (N). For "Total number of AEs" rows, multiple occurrences of the same AE are counted separately. For the frequency counts by preferred term, multiple occurrences of the same AE in one individual are counted only once.

For AE016SP, flag grade 4 events with "\*".

## ID: AE021SP

Adverse Events by Highest NCI CTCAE Grade STREAM Template: AET04

Analysis Population: Safety Evaluable Population

Analysis Variables: See mockup.

Include all AEs with an onset from first dose of study treatment through common closeout date

**Statistics and Calculation Methods**: Percentages are based on the number of patients in SE population (N). Multiple occurrences of the same AE in one individual are counted once at the greatest intensity/highest grade for this preferred term.

**Sort by:** Sort alphabetically by SOC, then within a SOC, sort by decreasing frequency of PT.

Numeric Precision and Formatting of Statistics: See mockup.

| MedDRA System Organ Class<br>MedDRA Preferred Term | Grade | Dose 1<br>(N=14) | Dose 2<br>(N=6) | All Patients<br>(N=20) |
|---|---|---|---|---|
| - Any adverse events - | any | 14 (100.0%) | 6 (100.0%) | 20 (100.0%) |
| | 5 | 2 ( 14.3%) | 1 ( 16.7%) | 3 ( 15.0%) |
| | 4 | 2 ( 14.3%) | 1 ( 16.7%) | 3 ( 15.0%) |
| | 3 | 4 ( 28.6%) | 4 ( 66.7%) | 8 ( 40.0%) |
| | 2 | 4 ( 28.6%) | 0 | 4 ( 20.0%) |
| | 1 | 2 ( 14.3%) | 0 | 2 ( 10.0%) |
| GASTROINTESTINAL DISORDERS | | | | |
| - Overall - | any | 13 ( 92.9%) | 6 (100.0%) | 19 ( 95.0%) |
| | 3 | 2 ( 14.3%) | 0 | 2 ( 10.0%) |
| | 2 | 4 ( 28.6%) | 1 ( 16.7%) | 5 ( 25.0%) |
| | 1 | 7 ( 50.0%) | 5 ( 83.3%) | 12 ( 60.0%) |
| DIARRHOEA | any | 10 ( 71.4%) | 4 ( 66.7%) | 14 ( 70.0%) |
| | 3 | 1 ( 7.1%) | 0 | 1 ( 5.0%) |
| | 2 | 4 ( 28.6%) | 0 | 4 ( 20.0%) |
| | 1 | 5 ( 35.7%) | 4 ( 66.7%) | 9 ( 45.0%) |
| VOMITING | any | 9 ( 64.3%) | 3 ( 50.0%) | 12 ( 60.0%) |
| | 2 | 1 ( 7.1%) | 1 ( 16.7%) | 2 ( 10.0%) |
| | 1 | 8 ( 57.1%) | 2 ( 33.3%) | 10 ( 50.0%) |
| NAUSEA | any | 7 ( 50.0%) | 4 ( 66.7%) | 11 ( 55.0%) |
| | 2 | 1 ( 7.1%) | 1 ( 16.7%) | 2 ( 10.0%) |
| | 1 | 6 ( 42.9%) | 3 ( 50.0%) | 9 ( 45.0%) |
| DRY MOUTH | any | 2 ( 14.3%) | 1 ( 16.7%) | 3 ( 15.0%) |
| | 1 | 2 ( 14.3%) | 1 ( 16.7%) | 3 ( 15.0%) |
| RETCHING | any | 2 ( 14.3%) | 1 ( 16.7%) | 3 ( 15.0%) |
| | 1 | 2 ( 14.3%) | 1 ( 16.7%) | 3 ( 15.0%) |
| CONSTIPATION | any | 1 ( 7.1%) | 1 ( 16.7%) | 2 ( 10.0%) |
| | 1 | 1 ( 7.1%) | 1 ( 16.7%) | 2 ( 10.0%) |
| DYSPEPSIA | any | 1 ( 7.1%) | 1 ( 16.7%) | 2 ( 10.0%) |
| | 1 | 1 ( 7.1%) | 1 ( 16.7%) | 2 ( 10.0%) |
| ABDOMINAL PAIN | any | 1 ( 7.1%) | 0 | 1 ( 5.0%) |
| | 1 | 1 ( 7.1%) | 0 | 1 ( 5.0%) |

#### ID: AF022SP

Listing of Patients with Dose Modification or Interruption Due to Adverse Events during Remission Induction Phase and Overall **STREAM Template**: AEL02

Analysis Population: Safety Evaluable Population

Variables Displayed: Add a new column to AEL02 for "The start

date of AE leading to dose modification/interruption".

Numeric Precision and Formatting of Statistics: See mockup.

## ID: AE023SP

Non-Serious Adverse Events Reported in >= 5% of Patients

STREAM Template: EUDRAT01

Analysis Population: Safety Evaluable Population

**Analysis Variables:** 

This table will be used to fulfill EudraCT and clintrials.gov disclosure requirements. It summarizes, for each treatment group, the number of patients, and the number of events, for non-serious AEs occurring in  $\geq 5\%$  of patients. Results will be displayed by SOC and PT within each SOC. Number of events at the SOC level is not displayed.

**Statistics and Calculation Methods**: Percentages are based on N in column heading. For each preferred term, multiple occurrences of the same AE in an individual are counted only once for the number of patients, and counted separately for the number of events.

**Sort by:** Display the data alphabetically by SOC, and by PT alphabetically within a SOC.

Numeric Precision and Formatting of Statistics: See mockup.

| | rituximab<br>(N=98) | |
|---|---|---|
| MedDRA System Organ Class<br>MedDRA Preferred Term | Patients | Events |
| Total number of patients with at<br>least one non-serious adverse event<br>occurring at relative frequency >=5%<br>and number of events | 95 | 1742 |
| Blood And Lymphatic System Disorders<br>Anaemia<br>Leukopenia<br>Neutropenia<br>Thrombocytopenia | 21<br>10<br>32<br>11 | 34<br>17<br>58<br>22 |
| Eye Disorders<br>Lacrimation Increased<br>Vision Blurred | 9<br>5 | 9<br>5 |
| Gastrointestinal Disorders<br>Abdominal Pain<br>Abdominal Pain Upper<br>Diarrhoea<br>Dyspepsia | 17<br>9<br>54<br>14 | 27<br>13<br>123<br>16 |

NOTE: Number of events includes all occurrences.

Rituximab—F. Hoffmann-La Roche Ltd WA25615: DAP Module 2

47

# ID: AE023.2SE

Serious Adverse Events, Fatal SAEs and SAEs Related to Study Medication **STREAM Template**: EUDRAT02

Analysis Population: SE Population

Analysis Variables: See mockup.

This table will be used to fulfill EudraCT disclosure requirements. It summarizes, by treatment group, by SOC and preferred term, the following:

- Number of patients with serious adverse events (SAEs)
- Number of SAEs
- Number of patients with fatal SAEs
- Number of SAEs resulting in death (fatal)
- Number of SAEs related to study medication
- Number of SAEs related to study medication and resulting in death

Number of events at the SOC level is not displayed.

Statistics and Calculation Methods: Percentages are based on N in column headings. For each preferred term, multiple occurrences of the same AE (that meet the relevant filter) in an individual are counted only once for the number of patients, and counted separately for the number of events.

**Sort by:** Display the data alphabetically by SOC, and by PT alphabetically within a SOC.

NOTE: Number of events includes all occurrences.

| MedDRA System Organ Class<br>MedDRA Preferred Term | Patients<br>(All) | Event<br>s<br>(All) | Patients<br>(Fatal) | Events<br>(Fatal) | Events<br>(Related) | Events<br>(Fatal<br>and<br>Related) |
|---|---|---|---|---|---|---|
| Blood And Lymphatic System Disorders | | | | | | |
| Anaemia | nnn | nnn | nnn | nnn | nnn | nnn |
| Coagulopathy | nnn | nnn | nnn | nnn | nnn | nnn |
| Febrile Neutropenia | nnn | nnn | nnn | nnn | nnn | nnn |
| Cardiac Disorders | | | | | | |
| Acute Myocardial Infarction | nnn | nnn | nnn | nnn | nnn | nnn |
| Atrial Fibrillation | nnn | nnn | nnn | nnn | nnn | nnn |

NOTE: Number of events includes all occurrences.

#### ID: AE024SP

Common Adverse Events Reported in >= 10% of Patients during Remission Induction Phase and Overall

STREAM Template: None

Analysis Population: Safety Evaluable Population

Analysis Variables:

Table of AEs grouped by System Organ Class (SOC) and listed by Preferred Term (PT) that occurred at a frequency ≥10% for each phase.

Note: "with at least one AE " means "with at least one AE which occurred for >=10% of patients".

Numeric Precision and Formatting of Statistics: See mockup.

| MedDRA System Organ Class | RITUXIMAB<br>(N=25) |
|-----------------------------------------------|---------------------|
| Total number of patients with at least one AE | 24 (96.0%) |
| UPPER RESPIRATORY TRACT INFECTION | 11 (44.0%) |
| HEADACHE | 10 (40.0%) |
| DIARRHOEA | 8 (32.0%) |
| EPISTAXIS | 7 (28.0%) |
| ARTHRALGIA | 6 (24.0%) |
| CHEST PAIN | 5 (20.0%) |
| CONJUNCTIVITIS | 5 (20.0%) |
| COUGH | 5 (20.0%) |
| GRANULOMATOSIS WITH POLYANGIITIS | 5 (20.0%) |
| NAUSEA | 5 (20.0%) |
| PYREXIA | 5 (20.0%) |
| HYPOGAMMAGLOBULINAEMIA | 3 (12.0%) |
| MIGRAINE | 3 (12.0%) |
| NASOPHARYNGITIS | 3 (12.0%) |
| PHARYNGITIS | 3 (12.0%) |
| RHINITIS | 3 (12.0%) |
| TREMOR | 3 (12.0%) |
| URINARY TRACT INFECTION | 3 (12.0%) |
| VIRAL INFECTION | 3 (12.0%) |
| VOMITING | 3 (12.0%) |

Investigator text for AEs is coded using MedDRA version 20.1. Percentages are based on N.

Table includes only AEs occurring in >=10% of patients in at least one treatment group. For frequency counts by preferred term, multiple occurrences of the same AE in an individual are counted only once.

# 7. SAFETY LABORATORY ANALYSES

# 7.1 Safety Laboratory Analyses

Safety hematology and serum chemistry laboratory samples are taken during each planned study visit.

Treatment-emergent clinically relevant laboratory test abnormalities are to be reported as adverse events on the Adverse Event eCRF and so will be reported as AEs. This is required for planned samples taken at study visits and also for any unscheduled samples taken.

For hematology and chemistry parameters, following summaries will be produced:

- Descriptive summaries, including changes from baseline, of values at baseline and throughout the study.
- The number of patients with values outside the normal upper and lower limit at each visit.

# 7.2 Acute-phase Reactants

Samples for measurement of erythrocyte sedimentation rate and C-reactive protein are taken during each study visit for analysis by the site's local laboratory. The parameters values and their changes from baseline will be summarized descriptively by visit and study phase.

# 7.3 Immunologic and Antibody Assessments

B- and T-cell populations are measured at baseline and each subsequent visit.

Samples for measurement of IgA, IgG, IgM and total immunoglobulins are taken at screening, baseline and then at each visit from Month 1 onwards. These will be summarized descriptively by visit and study phase and as changes from baseline.

# 7.4 Laboratory Output Specifications

#### ID: LB001SP

Laboratory Test results and Change from Baseline by Visit STREAM Template: LBT01

Analysis Population: Safety Evaluable Population

**Analysis Variables:** Single output file with separate page for each lab parameter as required by the protocol. Create tables for:

- Hematology: hematocrit, hemoglobin, red blood cells and indices (mean corpuscular volume, mean cell hemoglobin, mean corpuscular hemoglobin concentration), white blood cells, absolute differential [neutrophils, lymphocytes, monocytes, basophils], and platelet counts
- <u>Serum chemistry</u>: ALT/SGPT, alkaline phosphatase, AST/SGOT, calcium, chloride, creatinine, glycosylated hemoglobin (HbA<sub>1c</sub>), phosphate, potassium, sodium, total bilirubin (direct and indirect will be performed if total bilirubin is greater than the ULN), total protein, urea, uric acid

Sort order for tables: alphabetical by lab test (within hematology and chemistry)

Statistics and Calculation Methods: Per standard display.

Analysis visits to include are: Baseline, Weeks 1 to 3, Months 1, 2, 4, 6, 12 and 18. Values at visits to include only patients for whom a baseline value is included.

Numeric Precision and Formatting of Statistics: See mockup

```
Laboratory Test: SGPT/ALT (U/L)
                          Rituximab
                            (N=25)
                                Change from
           Value at Visit
                                  Baseline
Visit
Baseline
           24
 Mean (SD) 25.54 (22.20)
 Q1 - Q3 (IQR) XX. Y
 Median
                 xx.x - xx.x (xx.x)
 Min - Max 7.0 - 79.0
Week 1
               21
 n 21 20
Mean (SD) 27.43 (21.50) 1.75 (12.47)
Median 17.00 4.00
                                    2.0
 Q1 - Q3 (IQR) xx.x - xx.x (xx.x) xx.x - xx.x (xx.x)
Min - Max 7.0 - 95.0 -34.0 - 19.0
```

#### ID: LB004SP

Laboratory Abnormalities by Visit and Baseline Status STREAM Template: None

Analysis Population: Safety Evaluable Population

**Mock format:** See below for specific example with 4 extra columns.

Analysis Variables: See LB001SP for parameters to be included

and the appropriate analysis visits.

**Statistics and Calculation Methods**: Use the normal ranges given within the data. For each lab test and visit, include the following rows:

(a) For Baseline, should have rows for Low, Normal, and High.

(Always display all 3, even if count is 0.)

(b) For Post-baseline visits, should have rows for

Low - Change from Baseline

Low - Sustained

Low - Baseline Missing

Normal

High - Change from Baseline

High - Sustained

High - Baseline Missing

For post-baseline visits, only display the "Low – Baseline Missing" and "High – Baseline Missing" rows when they have a non-zero count. For all other rows, always display, even if count is 0.

## ALB.BASE1, ALB.RANGEB1, ALB.RANGE

Analysis visits to include are: Baseline, Weeks 1 to 3, Months 1, 2, 4, 6, 12 and 18.

Percentages are based on n.

**Numeric Precision and Formatting of Statistics:** See mockup (although we have just the one treatment group) – noting request above for rows to be presented.

#### Key Laboratory Assessments with Values Outside the Normal Limits Safety-Evaluable Patients

| Lab Tost | Visit | | Placebo<br>(N=66) | Leb 37.5 ng<br>(N=64) | Leb 125 mg<br>(N=62) | Lab 250 mg<br>(N=66) | A11 Lob<br>(N=192) |
|---|---|---|---|---|---|---|---|
| Alanine Aminotransferase | Baseline | n<br>Normal<br>High | 59 (89.4%)<br>7 (10.6%) | 59 ( 92.2%)<br>5 ( 7.8%) | 62<br>53 ( 85.5%)<br>9 ( 14.5%) | 66<br>58 ( 87.9%)<br>8 ( 12.1%) | 192<br>170 (88.5%)<br>22 (11.5%) |
| | Wook 4 | n<br>Normal<br>High - Change from Baseline<br>High - Sustained | 55 ( 91.7%)<br>1 ( 1.7%)<br>4 ( 6.7%) | 53<br>51 ( 96.2%)<br>1 ( 1.9%)<br>1 ( 1.9%) | 55<br>51 (92.7%)<br>1 (1.8%)<br>3 (5.5%) | 55 (91.7%)<br>1 (1.7%)<br>4 (6.7%) | 168<br>157 ( 93.5%)<br>3 ( 1.8%)<br>8 ( 4.8%) |
| | Waak 8 | n<br>Mormal<br>High - Change from Baseline<br>High - Sustained | 52<br>48 ( 92.3%)<br>1 ( 1.9%)<br>3 ( 5.8%) | 52<br>50 (96.2%)<br>2 ( 3.8%)<br>( 0.0%) | 54<br>50 ( 92.6%)<br>1 ( 1.9%)<br>3 ( 5.6%) | 50<br>43 (86.0%)<br>3 (6.0%)<br>4 (8.0%) | 156<br>143 (91.76)<br>6 (3.86)<br>7 (4.56) |
| | Wook 12 | n<br>Normal<br>High - Change from Baseline<br>High - Sustained | 48<br>43 (89.6%)<br>1 (2.1%)<br>4 (8.3%) | 44<br>43 ( 97.7%)<br>1 ( 2.3%)<br>( 0.0%) | 43<br>41 ( 95.3%)<br>( 0.0%)<br>2 ( 4.7%) | 47<br>41 (87.2%)<br>4 (8.5%)<br>2 (4.3%) | 134<br>125 ( 93.3%)<br>5 ( 3.7%)<br>4 ( 3.0%) |
| | Wook 16 | n<br>Normal<br>High - Change from Baseline<br>High - Sustained | 43<br>38 (88.4%)<br>2 (4.7%)<br>3 (7.0%) | 41<br>40 ( 97.6%)<br>1 ( 2.4%)<br>( 0.0%) | 39 (100.0%)<br>( 0.0%)<br>( 0.0%) | 42<br>35 (83.3%)<br>3 (7.1%)<br>4 (9.5%) | 122<br>114 ( 93.4%)<br>4 ( 3.3%)<br>4 ( 3.3%) |
| | Wook 20 | n<br>Normal<br>High - Change from Baseline<br>High - Sustained | 37<br>32 ( 86.5%)<br>4 ( 10.8%)<br>1 ( 2.7%) | 36<br>33 ( 91.7%)<br>3 ( 8.3%)<br>( 0.0%) | 37<br>33 ( 89.2%)<br>3 ( 8.1%)<br>1 ( 2.7%) | 36<br>31 (86.1%)<br>3 (8.3%)<br>2 (5.6%) | 109<br>97 (89.0%)<br>9 (8.3%)<br>3 (2.8%) |

High: >ULN; Low: <LLN.

Low & Change from Baseline: Normal or high at baseline, but low post-baseline.

Low & Sustained: Low at baseline, and low post-baseline.

Normal: Normal at visit. High & Change from Baseline: Normal or low at baseline, but high post-baseline.

High & Sustained: High at baseline, and high post-baseline.

pgm(/allergy/ilr/gb27862/final/programs/t\_lab\_shift) Source: Biostatistics Database (LOCKED) Datasets ( asl alb )

: Generated 09JAN14 07:40 Page 1 of 66

#### ID: LB005SP

Laboratory Test Shift Table: Highest NCI CTCAE Grade Post-Baseline: [High / Low] Hematology **STREAM Template:** LBT14

Analysis Population: Safety Evaluable Population

Mock format: See mockup below.

Analysis Variables: See LB001SP for parameters to be included and

the appropriate analysis visits.

Include patients with a missing baseline value.

**Statistics and Calculation Methods**: Use CTCAE grades, as appropriate. Use all available post-baseline data, not just windowed (analysis visit) results.

Percentages are based on n.

**Numeric Precision and Formatting of Statistics:** See mockup (although we have just the one treatment group) – noting request above for rows to be presented.

## **Additional Outputs:**

A similar output will be provided for the following safety lab categories:

| ID | Lab Category |
|---------|--------------|
| LB006SP | Chemistry |
| LB007SP | Urinalysis |

# Absolute neutrophil count

| Post-baseline NCI-CTCAE<br>Grade | Baseline NCI-CTCAE Grade | Rituximab<br>(N = nnn) |
|---|---|---|
| 0 | Total (n) | nn |
| | 1 | nn (xx.x%) |
| | 2 | nn (xx.x%) |
| | 3 | nn (xx.x%) |
| | 4 | nn (xx.x%) |
| | Missing | nn (xx.x%) |
| 1 | Total (n) | nn |
| | 1 | nn (xx.x%) |
| | 2 | nn (xx.x%) |
| | 3 | nn (xx.x%) |
| | 4 | nn (xx.x%) |
| | Missing | nn (xx.x%) |

ID: LB004SP

Listing of Normal
Ranges for Laboratory
Tests

STREAM Template: None

Analysis Population: Safety Evaluable Population

Variables Displayed: Name of Lab test, Lab ranges Low-High under Lab Parameters (with unit), grouped by age and gender.

| Lab Test | Lower Lab Range Upper Lab Range | | | | Unit | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | / | Age | Gende | er | Α | ge | Gende | r | |
| | <12 | >=12 | Female | Male | <12 | >=12 | Female | Male | |
| <lab test=""></lab> | XX | XX | XX | XX | XX | xx | XX | XX | XX |
| | XX | XX | XX | XX | XX | xx | XX | XX | XX |
| | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | XX | XX | XX | XX | XX | XX | XX | XX | XX |

Numeric Precision and Formatting of Statistics: See mockup

| ID: LB004.1SP | STREAM Template: LBL02A |
|---|---|
| Listing of lab | Analysis Population: Safety Evaluable Population |
| aonomantes | Numeric Precision and Formatting of Statistics: Add a column for "date of first drug administration" to LBL02A. |



## 8. VITAL SIGNS OUTPUT SPECIFICATIONS

During treatment visits, vital signs (temperature, pulse and BP) are measured immediately prior to the infusion, then every 15 minutes during the infusion until one hour, followed by every 30 minutes until the end of the infusion; a further reading is taken at least one hour after completion of the infusion. These data will be summarized within each visit by planned assessment time-point and also as changes from the within-visit pre-infusion value.

Additionally, vital signs plus height and weight will be summarized descriptively by visit (using pre-infusion values when appropriate), including changes from the baseline pre-infusion value.

# 8.1 Vital Signs Output Specifications

| ID: VS001SP | STREAM Template: VST01 |
|---|---|
| Vital Sign Results and | Analysis Population: Safety Evaluable Population |
| Change from Pre-<br>infusion by Infusion | Column Variables: Value after infusion and Change from Pre-infusion. |
| Number in Remission<br>Induction Phase | Analysis Variables: Separate tables in one file for each of: pulse rate (display as "heart rate" in the output), systolic blood pressure, and diastolic blood pressure. Use pre-infusion values only. |
| | Include planned infusions (in the remission induction phase). |
| | <b>Statistics and Calculation Methods:</b> Time-points to include are: pre-infusion and 0.25, 0.5, 0.75, 1, 1.5, 2, 6 hours post-infusion. |
| | Numeric Precision and Formatting of Statistics: See mockup |

| Time-point Relative to Infusion Start | | Value at Time-point | Change from Pre-<br>infusion |
|---|---|---|---|
| Infusion 1 | | • | |
| Pre-infusion | n | nn | |
| | Mean (SD) | xxx.x (xx.x) | |
| | Median | XXX.X | |
| | Q1 – Q3 (IQR) | xx.x-xx.x(xx.x) | |
| | Min-Max | XXX.X-XXX.X | |
| 0.25 hours Post | n | nn | nn |
| | Mean (SD) | xxx.x (xx.x) | xxx.x (xx.x) |
| | Median | XXX.X | XXX.X |
| | Q1 - Q3 (IQR) | xx.x-xx.x(xx.x) | xx.x-xx.x(xx.x) |
| | Min-Max | XXX.X-XXX.X | XXX.X-XXX.X |
| Infusion 2 | | | |

ID: VS002SP S

Vital Sign Results and Change from Baseline

by Visit

STREAM Template: VST01

Analysis Population: Safety Evaluable Population

Column Variables: Value at visit and Change from Baseline.

Statistics and Calculation Methods: Analysis visits to include are:

Baseline, Weeks 1 to 3, Months 1, 2, 4, 6, 9, 12, 15 and 18.

Values at visits to include only patients for whom a baseline value is

included.

Numeric Precision and Formatting of Statistics: See mockup

| Visit | | Value at Visit | Change from<br>Baseline |
|------------------|---------------|-----------------|-------------------------|
| Day 1 (Baseline) | n | nn | |
| | Mean (SD) | xxx.x (xx.x) | |
| | Median | XXX.X | |
| | Q1 – Q3 (IQR) | xx.x-xx.x(xx.x) | |
| | Min-Max | XXX.X-XXX.X | |
| Week 1 | n | nn | nn |
| | Mean (SD) | xxx.x (xx.x) | xxx.x (xx.x) |
| | Median | xxx.x | XXX.X |
| | Q1 – Q3 (IQR) | xx.x-xx.x(xx.x) | xx.x-xx.x(xx.x) |
| | Min-Max | XXX.X-XXX.X | XXX.X-XXX.X |
| Week 2 | n | nn | nn |
| | Mean (SD) | xxx.x (xx.x) | xxx.x (xx.x) |
| | Median | XXX.X | XXX.X |
| | Q1 – Q3 (IQR) | xx.x-xx.x(xx.x) | xx.x-xx.x(xx.x) |
| | Min-Max | XXX.X-XXX.X | XXX.X-XXX.X |

### ID: VS003SP

Vital Sign Results and Changes from Baseline Above and Below Specified Limits by Visit STREAM Template: None

Analysis Population: Safety Evaluable Population

**Analysis Variables:** Separate tables in one file for each of: pulse rate (display as "heart rate" in the output), systolic blood pressure, and diastolic blood pressure.

**Statistics and Calculation Methods:** Use pre-infusion values only. Analysis visits to include are: Baseline, Weeks 1 to 3, Months 1, 2, 4, 6, 9, 12, 15 and 18. Values at visits to include only patients for whom a baseline value is included.

Cut-off for each of the vital sign parameters are as follows:

| | | Value at Visit | | Change from Baseline | |
|---|---|---|---|---|---|
| Vital Sign | Units | Low | High | Decrease | Increase |
| Pulse rate | beats/min | < 50 | > 100 | ≥20 | ≥20 |
| Systolic blood pressure | mmHg | ≤90 | ≥140 | ≥ 20 | ≥20 |
| Diastolic blood pressure | mmHg | ≤50 | ≥90 | ≥ 15 | ≥15 |

As well as by-visit summaries, also summarise the number of patients who are low or high, or have a decrease/increase, at any post-baseline time-point. This will include <u>all</u> post-baseline data included in this analysis. A patient may count at most once towards the count on none, one or more of the 4 categories (see mockup).

Percentages are based on n.

Numeric Precision and Formatting of Statistics: See mockup

| Visit | | Rituximab<br>(N = nnn) |
|-------------------------|--------------|------------------------|
| Day 1 (Baseline) | n | nn |
| Value at Visit | <50 | nn (xx.x%) |
| | ≥50 to ≤100 | nn (xx.x%) |
| | >100 | nn (xx.x%) |
| Week 1 | n | nn |
| Value at Visit | <50 | nn (xx.x%) |
| | ≥50 to ≤100 | nn (xx.x%) |
| | >100 | nn (xx.x%) |
| Change from Baseline | Decrease ≥20 | nn (xx.x%) |
| | Increase ≥20 | nn (xx.x%) |
| Month 6 | n | nn |
| Value at ∀isit | <50 | nn (xx.x%) |
| | | , , |
| Change from Baseline | | |
| Any Post-baseline Value | n | nn |
| Values at Visits | <50 | nn (xx.x%) |
| | >100 | nn (xx.x%) |
| Changes from Baseline | Decrease ≥20 | nn (xx.x%) |
| | Increase ≥20 | nn (xx.x%) |

ID: VS004SP

Listing of Vital Sign Abnormalities STREAM Template: LBL02A\* (see mock)

Analysis Population: Safety Evaluable Population

**Numeric Precision and Formatting of Statistics:** See mockup Include patients with at least one post-baseline "abnormal" VS test.

Flag high (H) and low (L) results.

| Vital Sign Test<br>(Unit) | Center /<br>Patient ID | Age/Sex | Study<br>Day | Date | Result | Normal<br>Range |
|---|---|---|---|---|---|---|
| <∀ital Sign | | | | | | |
| Test> ( <unit>)</unit> | xxxx/xxx | XX | XX | ddMMMYY | xx L | XX-XX |
| | xxxx/xxx | xx | XX | ddMMMYY | xx L | xx-xx |
| | xxxx/xxx | xx | XX | ddMMMYY | xx H | XX-XX |
| | xxxx/xxx | xx | XX | ddMMMYY | xx | xx-xx |
| | xxxx/xxx | xx | XX | ddMMMYY | xx L | XX-XX |
| | xxxx/xxx | xx | XX | ddMMMYY | xx | xx-xx |
| | xxxx/xxx | XX | XX | ddMMMYY | хх Н | XX-XX |





# 9.1 Efficacy Output Specifications








































































Rituximab—F. Hoffmann-La Roche Ltd WA25615: DAP Module 2







Rituximab—F. Hoffmann-La Roche Ltd WA25615: DAP Module 2







## Appendix 1 Study Design



## Appendix 2 Schedule of Assessments

| | | | We | ek | | | | | N | /lonth | | Follow-Up | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | | Every 3<br>Months<br>after | | Extended |
| Visit <sup>a</sup> | Screen b | BL <sup>c</sup> | 1 | 2 | 3 | 1 | 2 | 4 | 6 | 9 | 12 | 15 | 18 | Month 18 d | WD | Follow-Up <sup>e</sup> |
| Day | | 1 | 8 | 15 | 22 | 29 | 60 | 120 | 180 | 270 | 365 | 455 | 545 | | | |
| Medications | | | | | | | | | | | | | | | | |
| Glucocorticoids IV f | | Х | | | | | | | | | | | | | | |
| Glucocorticoids PO g | | Х | Х | Х | х | Х | Х | х | Х | Х | Х | х | х | х | Х | Х |
| Pre-infusion medications h | | Х | Х | Х | Х | | | | | | | | | | | |
| Rituximab IV infusion | | Х | Х | Х | Х | | | | | | | | | | | |
| General Assessments | | | | | | | | | | | | | | | | |
| Informed Consent/<br>Child's Assent | х | | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | Х | | | | | | | | | | | | | | | |
| _ | | | | | | | | | | | | | | | | |
| Medical history | х | | | | | | | | | | | | | | | |
| Pregnancy test (serum) <sup>i</sup> | х | | | | | | | | | | | | | | | |
| Pregnancy test<br>(urine) <sup>i</sup> | | х | х | х | х | х | х | х | х | х | х | х | х | х | х | |
| 12-Lead ECG <sup>j</sup> | Х | | | | | | | | | | | | | | | |
| Height | Х | Х | | | | Х | Х | Х | Х | х | х | Х | Х | х | Х | х |
| Weight | Х | х | | | | Х | Х | Х | Х | х | х | Х | Х | X | х | X |
| Vital signs (pulse rate, systolic and diastolic blood pressure, and temperature) | х | x <sup>k</sup> | x <sup>k</sup> | x <sup>k</sup> | x <sup>k</sup> | х | х | х | х | х | х | х | x | х | х | х |

## Appendix 2 Schedule of Assessments (cont.)

| | | | | | | | N | lonth | | Follow-Up | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | | Every<br>3 Months<br>after | | Extended |
| Visit <sup>a</sup> | Screen b | BL° | 1 | 2 | 3 | 1 | 2 | 4 | 6 | 9 | 12 | 15 | 18 | Month 18 d | WD | Follow-Up <sup>e</sup> |
| Day | | 1 | 8 | 15 | 22 | 29 | 60 | 120 | 180 | 270 | 365 | 455 | 545 | | | |
| General Assessments (cont'd) | | | | | | | | | | | | | | | | |
| Physical examination | х | Х | х | х | х | х | х | Х | Х | Х | Х | Х | Х | x | Х | х |
| Chest X-ray <sup>1</sup> or CT scan <sup>m</sup> | Х | | | | | | | | | | | | | | Х | |
| Safety Assessments | | | | | | | | | | | | | | | | |
| Adverse events | | Х | х | х | х | х | х | Х | Х | Х | Х | х | Х | х | Х | х |
| Concomitant medications | X <sup>n</sup> | Х | х | х | х | х | х | Х | Х | Х | Х | Х | Х | х | Х | х |
| | | | Е | fficac | y Asse | essme | nts | | | | | | | | | |
| | | Ac | ute-Pl | hase I | Reacta | nt Ass | sessm | ents | | | | | | | | |
| C-reactive protein | х | Х | х | х | х | х | х | Х | х | х | Х | х | Х | х | Х | Х |
| Erythrocyte sedimentation rate | х | х | х | х | х | х | х | х | х | Х | Х | Х | Х | x | x | x |

1518

## Appendix 2 Schedule of Assessments (cont.)

| | | | | | | | | | | • | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Week Month Follow-U | | | | | | | | | Follow-Up | | | | |
| Visit <sup>a</sup> | Screen <sup>b</sup> | BL ° | 1 | 2 | 3 | 1 | 2 | 4 | 6 | 9 | 12 | 15 | 18 | Every<br>3 Months<br>after<br>Month 18 <sup>d</sup> | WD | Extended<br>Follow-Up <sup>e</sup> |
| Day | | 1 | 8 | 15 | 22 | 29 | 60 | 120 | 180 | 270 | 365 | 455 | 545 | | | |
| | | | La | borato | ory Ass | sessm | ents | | | | | | | | | |
| Hematology (CBC) | х | Х | х | х | х | х | х | х | Х | Х | Х | х | х | х | Х | х |
| Serum chemistry | х | Х | х | х | х | х | х | х | Х | Х | Х | Х | Х | х | Х | х |
| Urinalysis with microscopy and albumin to creatinine ratio | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | x |
| HbA <sub>1c</sub> s | | Х | | | | | х | Х | Х | Х | Х | Х | Х | х | Х | х |
| HBsAg, HBcAb, and HCV Ab and HBV DNA <sup>t</sup> | х | | | | | | | | | | | | | | | |
| Tuberculosis screening | х | | | | | | | | | | | | | | | |
| | | lmm | unolo | gic and | d Antik | ody A | ssess | ments | | | | | | | | |
| Immunoglobulins | х | Х | | | | х | х | Х | Х | Х | Х | х | Х | х | Х | х |
| CD19 B cells | | Х <sup>q</sup> | | Хq | | | | Х | Х | Х | Х | Х | Х | х | Х | х |
| FACS panel | | Х | х | х | х | х | х | Х | Х | Х | Х | х | Х | х | Х | х |
| Serum HACA sample | | Х | | | | | | Х | Х | Х | | | Х | x <sup>u</sup> | Х | x <sup>u</sup> |
| Serum ANCA sample v, w | х | | | | | х | | | Х | | Х | | Х | x <sup>u</sup> | Х | x <sup>u</sup> |
| | | | Pharr | nacok | inetic | Asses | sment | ts | | | | | | | | |
| Sample for rituximab levels | | x × | Хy | Хy | x× | х | х | х | х | х | | | х | x <sup>u</sup> | Х | x <sup>u</sup> |

ANCA = anti-neutrophil cytoplasmic antibody; CBC = complete blood count;

CT = computed tomography; ECG = electrocardiogram; eCRF = electronic Case Report Form; FACS = fluorescence-activated cell sorter; GFR = glomerular filtration rate; GPA = granulomatosis with polyangiitis; HbA<sub>1c</sub> = glycosylated hemoglobin; HBcAb = hepatitis B core antibody; HBsAg = hepatitis B surface antigen; HBV = hepatitis B virus; HCV Ab = hepatitis C virus antibodies; IV = intravenous; LLN = lower limit of normal; MPA = microscopic polyangiitis; PK = pharmacokinetic; PO = by mouth; PVDI = Pediatric Vasculitis Damage Index; WD = withdrawal.

- <sup>a</sup> For visit windows, please refer to protocol Appendix 2.
- b The screening visit must be completed within 28 days of the baseline visit.
- Assessments performed within 14 days of the baseline visit do not have to be repeated at the discretion of the investigator and if not clinically indicated.
- Until the common closeout date.

Rituximab—F. Hoffmann-La Roche Ltd WA25615: DAP Module 2

- e At the common closeout date, patients whose peripheral B cells remain depleted, will continue to attend study visits every 3 months until their peripheral B-cell counts have returned to pre-rituximab baseline levels or to within the normal range for the population, whichever is lower.
- Three times daily IV infusions of 30 mg/kg of methylprednisolone (up to 1 g/day, or equivalent) may be administered at any time, up to and including Day 1 (prior to the first rituximab infusion). If clinically indicated, and at the discretion of the investigator, an additional three daily doses of methylprednisolone (up to 1 g/day) can be given by IV infusion. No more than six doses in total can be given. All doses must be completed prior to the first rituximab infusion. The first rituximab infusion must occur no later than 14 days after the last dose of methylprednisolone infusion.
- g All patients will receive concomitant oral prednisolone or prednisone (1 mg/kg/day; up to 60 mg/day, or equivalent), which will be tapered to a minimum of 0.2 mg/kg/day (or 10 mg/day, whichever is lower) no later than Month 6.
- Patients should be premedicated with paracetamol/acetaminophen and cetirizine hydrochloride (or similar antihistamine), both according to labeled age-related doses, to be given 1 hour (±15 minutes) before each infusion of rituximab.
- To be completed for female patients of childbearing potential.
- After screening, only if clinically indicated.
- Vital signs should be taken immediately prior to infusion. During an infusion, record vital signs every 15 minutes for 1 hour; then every 30 minutes; and then at least 1 hour after the completion of the infusion.
- To be completed at screening and, if normal, only if indicated thereafter. If the chest X-ray is abnormal, repeat at Month 1 and as indicated thereafter.
- m CT scan to be completed only if indicated.
- Within the last 365 days of the screening visit.
  - CD19 B-cell samples to be obtained prior to infusion of rituximab.
- s Fasting is not required.
- After screening, only if clinically indicated.
- <sup>u</sup> After the Month 18 visit, samples should be taken every 6 months thereafter.
- ANCA testing performed at the screening visit to support a diagnosis of GPA or MPA may be performed locally or centrally. All other ANCA testing to be performed centrally.
- Also to be performed at time of flare.
- Y PK samples to be obtained prior to infusion of rituximab and 30 minutes following infusion of rituximab.
- PK samples to be obtained prior to infusion of rituximab.







